CLINICAL TRIAL: NCT03403881
Title: Avaliação de Uma intervenção de promoção Atividade física em Pacientes Com depressão Maior em Atendimento Ambulatorial (MOVEDEP): um Ensaio clínico Randomizado
Brief Title: Movement for Depression - An RCT Assessing the Effects of Physical Activity Promotion for People With MDD
Acronym: MOVEDEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0532
Record Dates: First submitted 2017-06-28; First posted 2018-01-19 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Major Depressive Disorder
Keywords: Exercise; Physical activity; Behavioral change; Depression; Major Depressive Disorder; Health promotion
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity promotion + TAU (Active Comparator): Physical activity promotion based on:
  * Pedometers use;
  * Weekly contact (telephone or face-to-face);
  * Contact based on a self-determination theory.
  TAU:
  Treatment as usual, which include medications. Medications were prescribed by psychiatrists not involved in the study participation.
  Interventions: Behavioral: Physical activity promotion + TAU
- Control (Placebo Comparator): Weekly calls with general health content.
  TAU:
  Treatment as usual, which include medications. Medications were prescribed by psychiatrists not involved in the study participation.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Physical activity promotion + TAU — Pedometer:
  Each patient will receive a pedometer with increasing weekly aims on number of steps during the trial.
  The number of steps to be achieved starts on 4.000 and increases progressively until the end of the trial.
  Behavioral strategy based on STD theory, and the assessment of barriers and facilitators of each patient.
  All patients were receiving treatment as usual
  Arms: Physical activity promotion + TAU
Behavioral: Control — Weekly call on general health aspects + treatment as usual
  Arms: Control

SUMMARY:
Randomized clinical trial that aims to increase physical activity levels in people with depression and to evaluate if the increase on PA levels has impact on clinical and biological measures.

DETAILED DESCRIPTION:
The contacts will be made by face-to-face interviews and telephone calls

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 65 years;
* diagnosis of Major Depressive Disorder (DSM-IV), assessed by a trained psychiatrist;
* score 7 or more in the HAM-D;
* do not present clinical comorbidities that limit or contra-indicate the practice of physical activity;
* be starting depression treatment at the Programa de transtorno do humor (PROTHUM) ;
* have acess to a computer and have a facebook account;
* be able to read and sign the consent term.

Exclusion Criteria:

* present other psychiatric diagnosis such as bipolar disorder, schizophrenia or use of alcohol or other drugs;
* be not liberated to the practice of physical exercises by the assistant psychiatrist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (blinded assessment) | At the end of the intervention (6 months)
  Hamilton scale for depressive symptoms assessed by a blinded psychiatrist. Clinician-administered semi-structured interview with 17 questions. It is designed to measure the severity of depressive symptoms in patients with a primary depressive illness. Higher scores means higher depressive symptoms. The cutoffs are the following: following severity ranges for the HAMD: no depression (0-7); mild depression (8-16); moderate depression (17-23); and severe depression (≥24). The maximum score is 52.

SECONDARY OUTCOMES:
Physical activity - self-report | At the end of the intervention (6 months)
  IPAQ
Physical activity levels - objective measure | At the end of the intervention (6 months)
  pedometer (only for intervention group)
Quality of life | At the end of the intervention (6 months)
  WHOQOL-BREF
Depressive symptoms (self-reported) | At the end of the intervention (6 months)
  Beck depressive inventory
Melancholia | At the end of the intervention (6 months)
  assessed using the CORE instrument
Weight | At the end of the intervention (6 months)
  Weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo B Fleck, PhD, Study Director — Researcher
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schuch FB, Vasconcelos-Moreno MP, Borowsky C, Zimmermann AB, Rocha NS, Fleck MP. Exercise and severe major depression: effect on symptom severity and quality of life at discharge in an inpatient cohort. J Psychiatr Res. 2015 Feb;61:25-32. doi: 10.1016/j.jpsychires.2014.11.005. Epub 2014 Nov 21. PMID 25439084
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Ward PB, Richards J, Ussher M, Schuch FB. Challenges Establishing the Efficacy of Exercise as an Antidepressant Treatment: A Systematic Review and Meta-Analysis of Control Group Responses in Exercise Randomised Controlled Trials. Sports Med. 2016 May;46(5):699-713. doi: 10.1007/s40279-015-0441-5. PMID 26707338
- [Background] Schuch FB, Vancampfort D, Richards J, Rosenbaum S, Ward PB, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. J Psychiatr Res. 2016 Jun;77:42-51. doi: 10.1016/j.jpsychires.2016.02.023. Epub 2016 Mar 4. PMID 26978184